CLINICAL TRIAL: NCT03275961
Title: Stress Management and Resiliency Training (SMART) Integrated Into Comprehensive Treatment of Major Depression: A Feasibility Study
Brief Title: Stress Management and Resiliency Training (SMART) Integrated Into Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ashok Seshadri, Consultant, Instructor in Psychiatry, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-007944
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressed Subjects (Experimental): Subjects will undergo an 8 week behavioral program with Stress Management and Resiliency Training.
  Interventions: Behavioral: Stress Management and Resiliency Training

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training — Subjects will undergo an 8 week behavioral program. Treatment will consist of weekly group therapy sessions in small groups with core practices to apply the principles of SMART.
  Other Names: SMART

SUMMARY:
The investigators are doing this research study to find out if the Stress Management and Resiliency Training (SMART) therapy will help subjects with their major depression treatment.

DETAILED DESCRIPTION:
The investigators propose to conduct an initial feasibility study in a sample of patients in treatment for major depression using SMART. The intervention will be weekly group therapy session of SMART for 8 weeks duration. Once enrolled, participants will complete a Structured Clinical Interview for Diagnosis (SCID). The SCID will primarily serve to confirm a diagnosis of Major Depressive Disorder. Each study intervention group (3-4 groups) will be composed of 6-8 research participants per group. There will be no comparison group. The investigators aim to assess adherence with goal of 75% completion of the 8 sessions of SMART and of the homework assignments. Resilience will be measured with the Connor-Davidson resilience scale. Secondary outcomes will include subjective and objective clinical rating scales for major depression.

ELIGIBILITY:
Inclusion Criteria:

* Attending the Mayo Clinic Depression Center and Behavioral Health Clinic at Mayo Clinic Health System, Austin, Minnesota
* DSM-V diagnostic confirmation of major depressive disorder (MDD)
* Baseline PHQ-9 scores in the range of ≥6-≤19, and HAMD-17 score 8-18, or QIDS-C16 score of 6-20
* Able to speak English
* Participants will continue taking any prescribed medications from their clinical treatment team
* Patients with co-morbid secondary diagnoses of persistent depressive disorder and generalized anxiety disorders will be included in the study.

Exclusion Criteria:

* Participants with bipolar disorder
* Active psychosis
* Active suicidal ideations
* Active substance abuse meeting criteria for substance use disorders except nicotine
* Obsessive compulsive disorder
* Active Panic disorder with agoraphobia, other phobic disorder
* Active Posttraumatic stress disorder
* Active Severe personality disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Connor-Davidson Resilience Scale Score | baseline, 8 weeks
  The Connor-Davidson Resilience Scale (CD-RISC), a 25-item scale, was developed to measure resiliency. CD-RISC has been evaluated and has been found to have good internal consistency (α = .89), test-retest reliability (intraclass correlation coefficient = .87), and positive correlation with multiple related measures with ability to distinguish between participants with lesser and greater resilience. The scores can range from 0 to 100. The mean score in a general population sample was 80.7 and in psychiatric outpatients 68. A positive change with increasing scores will indicate improvement in resilience.

SECONDARY OUTCOMES:
Change in Hamilton Rating Scale for Depression Score | baseline, 8 weeks
  The Hamilton Rating Scale for Depression (HAMD-17) is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. The 17 items are rated on either a 5-point (0-4) or a 3-point (0-2) scale. In general, the 5 point scale items use a rating of 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. The 3-point scale items use a rating of 0=absent; 1=probable or mild; 2=definite. The total HAMD-17 score ranges from 0 (not ill) to 52 (severely ill). A negative change indicates improvement in the subject's depression/anxiety symptoms, and a positive change indicates a worsening of the subject's depression/anxiety symptoms.
Change in Patient Health Questionnaire-9 Score | baseline, 8 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered 9-item scale which scores each of the 9 DSM-V criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 6-10,11-15, 16-20, and >20 represented mild, moderate, moderately severe, and severe depression, respectively.
Change in Quick Inventory of Depressive Symptoms Score | baseline, 8 weeks
  The 16-item Quick Inventory of Depressive Symptomatology (QIDS) designed to assess the severity of depressive symptoms. The QIDS assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) to diagnose a major depressive episode. The scores can range from 0 to 27, with 0 being no depression to 27 being very severe depression. Increasing scores indicate worsening depression and decreasing scores indicate improving depression.
Change in Generalized Anxiety Disorder-7 Score | baseline, 8 weeks
  Generalized Anxiety Disorder 7 (GAD-7) is a 7 item self-report scale which scores the symptoms of generalized anxiety disorder (GAD) from "0"( not at all) to "3"( nearly every day). Cut points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety on the GAD-7.
Change in Perceived Stress Scale Score | baseline, 8 weeks
  The Perceived Stress Scale is a 10 item self-administered scale that measures the degree to which one's life are appraised as stressful. The scores can range from 0( no stress) to 40( very high stress). Scores between 0-13 are considered low stress, 14-26- moderate stress and 27-40- high stress. A decreasing trend of scores would indicate improvement in perceived stress levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Seshadri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seshadri A, Clark MM, Kung S, Fuller-Tyszkiewicz M, Sood A, Dammen KC, Rico JA, Tye SJ, McGillivray J, Frye MA. Feasibility Study of Stress Management and Resiliency Training (SMART) in Patients With Major Depressive Disorder. Prim Care Companion CNS Disord. 2020 Apr 30;22(3):19m02556. doi: 10.4088/PCC.19m02556. PMID 32369689